CLINICAL TRIAL: NCT05388448
Title: A Phase 2 Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of Sanfetrinem Cilexetil Administered Orally to Adults With Newly Diagnosed, Smear-Positive, Rifampicin-Susceptible Pulmonary Tuberculosis
Brief Title: EBA, Safety and Tolerability of Sanfetrinem Cilexetil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Collaborators: GlaxoSmithKline (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TASK-009-SANF
Record Dates: First submitted 2022-01-25; First posted 2022-05-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: tuberculosis; early bactericidal activity; bedaquiline; delamanid
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — sanfetrinem cilexetil; Rifampin

STUDY DESIGN:
Intervention Model Description: Approximately 51 participants (3 groups of approximately 15 participants receiving IP including replacements in Stage 1) will be enrolled. 26 participants were enrolled in stage 1 and 25 are planned to be enrolled in stage 2. Participants will be between 18 and 65 years old (inclusive), with newly diagnosed, smear or Xpert MTB/RIF-positive, rifampicin susceptible pulmonary TB.
Masking Description: Laboratory personnel are blinded to treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sanfetrinem cilexetil 1.6 gram 12 hourly (Experimental): Sanfetrinem cilexetil 1.6g will be given orally 12 hourly for 14 consecutive days.
  Interventions: Drug: Sanfetrinem Cilexetil
- Rifampicin 35 mg/kg once daily (Experimental): Rifampicin 35 mg/kg will be given orally once daily for 14 consecutive days.
  Interventions: Drug: Rifampicin
- Sanfetrinem cilexetil 2.4 gram once daily (Experimental): Sanfetrinem cilexetil 2.4 g will be given orally daily for 14 consecutive days.
  Interventions: Drug: Sanfetrinem Cilexetil

INTERVENTIONS:
Drug: Sanfetrinem Cilexetil — Sanfetrinem cilexetil powder, weighed for dose and administered as a suspension in water.
  Amx/CA 250/125 mg tablets Rifampicin 150 mg, 300 mg and 600 mg tablets or capsules
  Other Names: Compound number GV118819
  Arms: Sanfetrinem cilexetil 1.6 gram 12 hourly; Sanfetrinem cilexetil 2.4 gram once daily
Drug: Rifampicin — Rifampicin will be administered at a dose of 35 mg/kg once daily for 14 days with or without sanfetrinem cilexetil.
  Other Names: Rifadin
  Arms: Rifampicin 35 mg/kg once daily

SUMMARY:
To evaluate the 2-week bactericidal activity, pharmacokinetics, safety and tolerability of sanfetrinem cilexetil in participants with rifampicin-susceptible pulmonary tuberculosis.

DETAILED DESCRIPTION:
A single-centre, open-label, clinical trial in two stages. Stage 1 will recruit 20 participants followed by a recruitment pause and an interim analysis to determine if sanfetrinem cilexetil has early bactericidal activity (EBA). Should EBA be demonstrated, stage 2 will focus on optimising sanfetrinem cilexetil.

All treatments will be administered orally (PO) on days 1-14. The treatments are:

Stage 1:

* Sanfetrinem cilexetil 1.6 g PO 12-hourly
* Rifampicin 35 mg/kg PO once daily (OD)*

An interim analysis is planned after stage 1 to review the pharmacokinetics (PK), safety, tolerability and EBA of sanfetrinem cilexetil. Results of stage 1 will determine whether stage 2 should proceed and if any modifications in dose, duration or combinations are required for Stage 2. If deemed possible, a PK-EBA model will be derived using only stage 1 from which clinical trial simulations will be conducted to inform the design of stage 2. If EBA is not demonstrated, the study will be stopped after stage 1.

Stage 2:

* Rifampicin 35 mg/kg po OD*
* Sanfetrinem cilexetil 2.4 g PO OD

Five of the rifampicin 35 mg/kg arm participants will be recruited in stage 1 and the remainder in stage 2.

Participants on rifampicin will serve as control for the EBA quantitative mycobacteriology.

The study will not be blinded but the mycobacteriology laboratory staff performing the endpoint assays will remain blinded until analysis of the EBA results.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to meet all of the following criteria in order to be randomized.

  1. Provide written, informed consent prior to all trial-related procedures.
  2. Male or female, aged between 18 and 65 years, inclusive.
  3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
  4. Newly diagnosed, previously untreated, rifampicin-susceptible pulmonary TB.
  5. A chest X-ray picture taken at screening which, in the opinion of the investigator, is consistent with TB.
  6. Sputum positive on direct microscopy for acid-fast bacilli on at least one sputum sample (at least 1+ on the IUATLD/WHO scale) or GeneXpert cycle threshold of medium or high.
  7. Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 ml or more).
  8. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

Female participant/ female sexual partner - bilateral oophorectomy

* bilateral tubal ligation
* hysterectomy
* postmenopausal with no menses for at least 12 consecutive months Male participant/ male sexual partner - vasectomy
* bilateral orchidectomy more than three months prior to screening

Effective birth control methods:

1. Participant is not heterosexually active or practicing sexual abstinence
2. Double barrier method which can include a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); or
3. Barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner.

Exclusion Criteria:

* Participants will be excluded from participation if they fulfil any of the following criteria.

  1. Evidence of clinically significant conditions or findings, other than TB, that might compromise safety or the interpretation of trial endpoints, per discretion of the investigator.
  2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the investigator.
  3. Clinically significant evidence of extrathoracic TB, as judged by the investigator.
  4. History of allergy to any of the trial IP/s or related substances i.e. β-lactams and penicillin, as confirmed by the clinical judgement of the investigator.
  5. Alcohol or drug abuse, that in the opinion of the investigator, is sufficient to compromise the safety or cooperation of the participant.
  6. HIV positive ONLY IF:

     * CD4 < 250cells/mm3
     * On ART
  7. Participation in other clinical studies with investigational agents within 8 weeks prior to trial start (with the exception of COVID-19 vaccines).
  8. Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of trial participation. Male participant planning to conceive a child within the anticipated period of participating in the trial.
  9. Treatment received with any drug active against M.tb (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides), or with immunosuppressive medications such as TNF-alpha inhibitors within 2 weeks prior to screening, or systemic corticosteroids for more than 7 days within 2 weeks prior to screening.
  10. Participants with the following toxicities at screening as defined by the enhanced CTCEA toxicity table

      1. creatinine >1.5 times upper limit of normal [ULN];
      2. haemoglobin <8.0 g/dL;
      3. platelets <50x109 cells/L;
      4. serum potassium <3.0 mmol/L;
      5. aspartate aminotransferase (AST) ≥3.0 x ULN;
      6. alanine aminotransferase (ALT) ≥3.0 x ULN;
      7. Total white cell count <1.5 cells/L
  11. For participants undergoing PET/CT, the following are excluded:

      1. Participants with diabetes (Type 1 or 2) with point of care HbA1c above 6.5, or random glucose over 11.1 mmol/L.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Rate of change in mycobacterium tuberculosis (Mtb) load in sputum from pre-treatment to Day 14 on-treatment, based on colony forming unit (CFU) count on solid culture media (7H11 agar plates) | 14 days
  Early bactericidal activity (EBA) will be determined, per treatment arm, as the rate of change in log10 CFU count per ml sputum over the treatment period day 0 to day 14, and described using linear, bi-linear or non-linear regression of log10CFU count over time and relation to drug exposure.

SECONDARY OUTCOMES:
Rate of change in mycobacterium tuberculosis (Mtb) load in sputum from pre-treatment to Day 14 on-treatment, based on time to positive (TTP) culture in the BACTEC MGIT 960 liquid culture system | 14 days
  EBA will be determined, per treatment arm, by the rate of change in time to culture positivity (TTP) over the treatment period day 0 to day 14, and described using linear, bi-linear or non-linear regression of TTD over time and relation to drug exposure
Number of patients with abnormal safety and tolerability findings following the study regimens, administered for 14 days | 14 days
  The pooled incidence of the following events will be summarized by treatment group for further analysis:
  Incidence of treatment-emergent adverse events (TEAEs); Incidence of TEAEs by Severity; Incidence of drug related TEAEs; Incidence of Serious TEAEs; Incidence of TEAEs leading to early withdrawal; Incidence of TEAEs leading to death Incidence of treatment-emergent adverse events (TEAEs); Incidence of TEAEs by Severity; Incidence of drug related TEAEs; Incidence of Serious TEAEs; Incidence of TEAEs leading to early withdrawal; Incidence of TEAEs leading to death

CONTACTS AND LOCATIONS:
Locations (1):
- TASK Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramon-Garcia S, Gonzalez Del Rio R, Arenaz-Callao MP, Boshoff HI, Rullas J, Anca S, Cacho Izquierdo M, Porras de Francisco E, Perez Herran E, Santos-Villarejo A, Mendoza-Losana A, Ferrer-Bazaga S, Thompson CJ, Barros Aguirre D, Bates RH. Sanfetrinem, an oral beta-lactam antibiotic repurposed for the treatment of tuberculosis. Drug Resist Updat. 2025 May;80:101213. doi: 10.1016/j.drup.2025.101213. Epub 2025 Feb 15. PMID 40020440
- [Derived] Ramon-Garcia S, Del Rio RG, Arenaz-Callao MP, Boshoff H, Rullas J, Anca S, Izquierdo MC, de Francisco EP, Herran EP, Santos-Villarejo A, Mendoza-Losana A, Ferrer-Bazaga S, Thompson CJ, Aguirre DB, Bates RH. Sanfetrinem, an oral beta-lactam antibiotic repurposed for the treatment of tuberculosis. bioRxiv [Preprint]. 2024 Oct 10:2024.10.10.617558. doi: 10.1101/2024.10.10.617558. PMID 39803560
- See also: TASK Homepage - clinical research institute and social enterprise — http://www.task.org.za/